CLINICAL TRIAL: NCT05446506
Title: Comparative Study for Serum Levels of Otolin-1 and Vitamin D in pre-and Post-treatments of Patients With Benign Paroxysmal Positional Vertigo
Brief Title: Serum Levels of Otolin-1 and Vitamin D in Pre- and Post-treatments of BPPV
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Suwicha Isaradisaikul Kaewsiri, Clinical Professor, Department of Otolaryngology, Chiang Mai University
Other Study IDs: ENT-2563-07658
Record Dates: First submitted 2022-04-12; First posted 2022-07-06 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: otolin-1; vitamin D; biomarker; inner ear
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BPPV is the most common cause of vertigo. The pathophysiology of BPPV has not been cleared, several studies show that symptoms are caused by the displacement of otoconia from the macula of the utricle into the semicircular canals. These calcium carbonate particles then stimulate non-physiological movement of the endolymph leading to a false sensation of angular acceleration.

Biomarkers represent measurable products of biological processes, thus making an assessment of those processes more practical. Biomarkers in circulation are powerful indicators of normal and pathological biological processes, as well as, responses to pharmacological treatments. The inner ear-inclusive protein that has been published included Otolin-1, Otoconin-90/95, Prestin, Otoancorin, Otogelin, α-tectorin, β-tectorin and Cochlin.

DETAILED DESCRIPTION:
The posterior canal BPPV is the most common BPPV variant, diagnosed with the Dix-Hallpike test. The lateral canal BPPV is diagnosed with a supine roll test. After treatment of the posterior canal BPPV with a single cycle of the CRP, the rate of negative DHT was 68-80% in the 1st week. Rate of an absence of vertigo and nystagmus on the supine roll test after-treatment of the lateral canal BPPV with the barbecue maneuver plus forced prolonged positioning was 81%.

Biomarkers are often measured in body fluids, they eliminate the need for costly modalities to diagnose and monitor progression. Otolin-1 is a secreted glycoprotein whose messenger RNA (mRNA) expression is restricted to the inner ear, specifically the support cells of the vestibular maculae, semicircular canal cristae, organ of Corti, and marginal cells of the stria vascularis. Otolin-1 blood levels are significantly higher in patients older than 65 years old and increased prevalence of BPPV with age. There were reports of a relationship between vitamin D and otolin-1. Significantly higher serum levels of the otolin-1 protein in patients with BPPV than in healthy controls has been reported. This also confirmed evidence of the otolin-1 as a potential biomarker for BPPV episodes and maybe clinically used to promote better management of BPPV. No data on inner ear biomarkers has been exited in Thailand.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80 years
2. History of brief episodes of positioning vertigo
3. Positive positioning test; either Dix-Hallpike test or supine roll test in one or both ears
4. First diagnosis of BPPV or recurrent BPPV

Exclusion Criteria:

1. Clinical symptoms or sign of other central or peripheral vestibular disorder
2. Previous history of balance disorders (for controlled group) or Previous history of balance disorders except BPPV (for BPPV group)
3. Active infection
4. Active cancer disease
5. Conditions that may affect the level of otolin-1 such as previous mastoidectomy
6. Conditions that may affect the level of vitamin D such as cardiovascular disease, diabetes mellitus type2, chronic liver disease, osteoporosis osteomalacia and active symptoms of migraine
7. Major health conditions; except common chronic conditions e.g. hypertension, hypothyroidism, hypercholesterolemia, and reflux
8. Major systemic illness, were undergoing active cancer treatment, took prednisone above 10 mg daily, took other immunosuppressive drugs, took any medications for rheumatoid arthritis other than NSAIDs, or had received antibiotics in the previous 6 months
9. Unable to complete Thai-Dizziness handicap inventory questionnaire
10. Unable to obtain the blood specimen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: BPPV cases in outpatient Ear Nose and Throat (ENT) Clinic at CMU Hospital, Faculty of Medicine, Chiang Mai University during the study period.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Level of serum otolin-1 and vitamin D | Day 0 and 7±3days after treatment
  changes of Level of serum otolin-1 and vitamin D before and after treatment of BPPV

SECONDARY OUTCOMES:
Correlation of serum otolin-1 and vitamin D | Day 0 and 7±3days after treatment
  Correlation of serum otolin-1 and vitamin D before and after treatment period in BPPV patients

CONTACTS AND LOCATIONS:
Overall Officials: Suwicha Kaewsiri, MD, Principal Investigator — Department of Otolaryngology , Faculty of Medicine, Chiang Mai University
Locations (1):
- Department of Otolaryngology Faculty of Medicine, Chiang Mai University 110 Intawaroros Road, Sriphum, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Parham K, Sacks D, Bixby C, Fall P. Inner ear protein as a biomarker in circulation? Otolaryngol Head Neck Surg. 2014 Dec;151(6):1038-40. doi: 10.1177/0194599814551127. Epub 2014 Sep 22. PMID 25245136
- [Result] Isaradisaikul S, Navacharoen N, Hanprasertpong C, Kangsanarak J, Panyathong R. Causes and time-course of vertigo in an ear, nose, and throat clinic. Eur Arch Otorhinolaryngol. 2010 Dec;267(12):1837-41. doi: 10.1007/s00405-010-1309-9. Epub 2010 Jun 22. PMID 20567978
- [Result] Lynn S, Pool A, Rose D, Brey R, Suman V. Randomized trial of the canalith repositioning procedure. Otolaryngol Head Neck Surg. 1995 Dec;113(6):712-20. doi: 10.1016/S0194-59989570010-2. PMID 7501382
- [Result] Burton MJ, Eby TL, Rosenfeld RM. Extracts from the Cochrane Library: modifications of the Epley (canalith repositioning) maneuver for posterior canal benign paroxysmal positional vertigo. Otolaryngol Head Neck Surg. 2012 Sep;147(3):407-11. doi: 10.1177/0194599812457134. Epub 2012 Aug 11. PMID 22886077
- [Result] Bhattacharyya N, Gubbels SP, Schwartz SR, Edlow JA, El-Kashlan H, Fife T, Holmberg JM, Mahoney K, Hollingsworth DB, Roberts R, Seidman MD, Prasaad Steiner RW, Tsai Do B, Voelker CC, Waguespack RW, Corrigan MD. Clinical Practice Guideline: Benign Paroxysmal Positional Vertigo (Update) Executive Summary. Otolaryngol Head Neck Surg. 2017 Mar;156(3):403-416. doi: 10.1177/0194599816689660. PMID 28248602
- [Result] Mulry E, Parham K. Inner Ear Proteins as Potential Biomarkers. Otol Neurotol. 2020 Feb;41(2):145-152. doi: 10.1097/MAO.0000000000002466. PMID 31789810
- [Result] Sacks D, Parham K. Preliminary Report on the Investigation of the Association Between BPPV and Osteoporosis Using Biomarkers. Otol Neurotol. 2015 Sep;36(9):1532-6. doi: 10.1097/MAO.0000000000000853. PMID 26375977
- [Result] Koestner A, Long JF. Ultrastructure of canine distemper virus in explant tissue cultures of canine cerebellum. Lab Invest. 1970 Aug;23(2):196-201. No abstract available. PMID 5464974
- [Result] Parham K, Kuchel GA, McElhaney JE, Haynes L. A Relationship Between Blood Levels of Otolin-1 and Vitamin D. Otol Neurotol. 2018 Apr;39(4):e269-e273. doi: 10.1097/MAO.0000000000001747. PMID 29533337
- [Result] Wu Y, Han W, Yan W, Lu X, Zhou M, Li L, Guan Q, Fan Z. Increased Otolin-1 in Serum as a Potential Biomarker for Idiopathic Benign Paroxysmal Positional Vertigo Episodes. Front Neurol. 2020 May 13;11:367. doi: 10.3389/fneur.2020.00367. eCollection 2020. PMID 32477244